CLINICAL TRIAL: NCT01509053
Title: Open-label Study to Assess Hospitalization Rates in Adult Schizophrenic Patients Treated With Oral Antipsychotics for 6 Months and IM Depot Aripiprazole for 6 Months, Respectively, in a Naturalistic Community Setting, Europe, Canada and Asia
Brief Title: Open-label Study to Compare Hospitalization Rates of Schizophrenic Patients Treated With Oral Antipsychotics Versus IM Depot Aripiprazole
Acronym: ARRIVE- EU
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 31-11-284
Record Dates: First submitted 2011-12-13; First posted 2012-01-12 (Estimated); Results first posted 2014-01-16 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-02

CONDITIONS: Schizophrenia
Keywords: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aripiprazole IM depot injection (Experimental): Patients who had no history of tolerability to oral aripiprazole received 10-15 mg/day (up to 30 mg/day) oral aripiprazole for 1 to 4 weeks to determine tolerability in the Tolerability Assessment Phase prior to receiving treatment with aripiprazole IM Depot. In the Open-label Aripiprazole IM Depot Phase, participants received aripiprazole intramuscular (IM) Depot 400 mg injection (dosage could be adjusted to 300 mg at the investigator's discretion) monthly in the clinic for a total of 6 injections + concomitant oral aripiprazole 10-15 mg/day for the first 14 days. Participants at the investigator's discretion were eligible to continue to receive aripiprazole IM depot (400 or 300 mg) injection monthly in the Open-label Aripiprazole IM Depot Extension phase. Oral aripiprazole was available as rescue medication if necessary.
  Interventions: Drug: Aripiprazole (Abilify®) IM Depot Injection; Drug: Oral aripiprazole

INTERVENTIONS:
Drug: Aripiprazole (Abilify®) IM Depot Injection — 400 mg IM depot injection every 26-30 days. Dosage may be adjusted at the investigator's discretion to 300 mg.
  Number of injections: 6. Participants have the option of entering the extension phase of the study and continuing with injections every 26-30 days until the drug is either commercially available, or December 2014.
  Other Names: ABILIFY®
Drug: Oral aripiprazole — Oral aripiprazole tablets 10-15 mg/day (up to 30 mg/day).

SUMMARY:
The purpose of this study is to compare retrospective hospitalization rates of schizophrenic patients treated with oral antipsychotics to prospective hospitalization rates of these patients treated with IM depot aripiprazole.

DETAILED DESCRIPTION:
Nonadherence to antipsychotic medications remains a frequent cause of relapse among patients with schizophrenia, increasing hospitalization rates, hospitalization days, and hospitalization costs. Among hospitalized adults, schizophrenia is the fourth most commonly diagnosed illness and has the seventh longest mean duration of hospital stay in the US. Frequent relapses and hospitalization can affect quality of life in these patients. Long-acting injections (intramuscular depot) antipsychotic medication is a means to treatment adherence and increased quality of life for patients with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are able to provide written informed consent. If the Institutional Review Board (IRB) requires consent by a legally acceptable representative in addition to the subject, all required consents must be obtained prior to any protocol-required procedure.
* Male and female subjects 18 to 65 years of age, inclusive
* Current diagnosis of schizophrenia as defined by Diagnostic and Statistical Manual of Mental Disorders (DSM-IV-TR) criteria and a history of the illness for at least 1 year (12 months)
* Subjects who in the investigator's judgment would benefit from extended treatment with a long-acting injectable formulation
* Subjects who have at least 1 inpatient psychiatric hospitalization in the 2 years (24 months) prior to screening, but have been managed as outpatients for the 4 weeks prior entering the study
* Subjects must have been on oral antipsychotic treatment for the full 7 months prior to the screening phase Subjects who have shown response to previous antipsychotic treatment.
* Subjects who understand the nature of the trial and are able to follow the protocol requirements.

Exclusion Criteria:

* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated), or have been incarcerated in the past 7 months for any reason must not be enrolled into this trial.
* Subjects who may require potent CYP2D6 or CYP3A4 inhibitors or CYP3A4 inducers during the trial.
* Any subject who requires or may need any other antipsychotic medications during the course of the trial, other than allowed rescue medication.
* Subjects who are known to be allergic, intolerant, or unresponsive to prior treatment with aripiprazole or other quinolinones.
* Subjects with a history of hypersensitivity to antipsychotic agents.
* Subjects deemed intolerant of receiving injectable treatment.
* Subjects who have received electroconvulsive therapy within the last 7 months prior to screening.
* Subjects with a history of neuroleptic malignant syndrome or clinically significant tardive dyskinesia as assessed by the investigator.
* Subjects with a current DSM-IV-TR diagnosis other than schizophrenia, including schizoaffective disorder, major depressive disorder, bipolar disorder, delirium, dementia, amnestic or other cognitive disorders. Also, subjects with borderline, paranoid, histrionic, schizotypal, schizoid, or antisocial personality disorder.
* Subjects requiring hospitalization for any psychiatric reason during the 4 weeks prior to signing the Informed Consent Form (ICF) or during the screening period.
* Subjects without at least 1 inpatient psychiatric hospitalization in the last 2 years (24 months) prior to screening.
* Subjects who have met DSM-IV-TR criteria for any significant substance use disorder within 3 months prior to screening.
* Subjects who are considered treatment-resistant to antipsychotic medication other than clozapine.
* Treatment with long-acting injectable antipsychotics in which the last dose was within 7 months prior to screening.
* Subjects who have not been treated with oral antipsychotics for 7 months prior to screening.
* Subjects who have a significant risk of committing suicide
* Subjects who have a history or evidence of a medical condition that would expose them to an undue risk of a significant adverse event or interfere with assessments of safety or efficacy during the course of the trial
* Sexually active males and females who will not commit to utilizing birth control during the trial and for up to 180 days following the trial.
* Abnormal laboratory or physical examination results indicating a condition which may interfere with the results of the study or pose a safety risk to the subject.
* Subjects who have previously enrolled in an aripiprazole IM depot clinical study or who have participated in any clinical trial with an investigational agent within the past 30 days.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-01; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim Peters-Strickland, Study Director — Otsuka Pharmaceutical Development & Commercialization, Inc.
Locations (10):
- Belgium (4):
  - Bruges
  - Brussels
  - Kortenberg
  - Liège
- Bulgaria (4):
  - Lovech
  - Novi Iskar
  - Pazardzhik
  - Tzerova Koria
- Canada (2):
  - Penticton, British Columbia
  - Chatham, Ontario

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study included a Tolerability Assessment Phase A (if applicable), an Open-Label Aripiprazole IM Depot Phase B and an Open-Label Aripiprazole IM Depot Extension Phase C.
Groups:
- Oral Aripiprazole Tablets and Aripiprazole IM Depot Injection: Patients who had no history of tolerability to oral aripiprazole received 10-15 mg/day (up to 30 mg/day) oral aripiprazole for 1 to 4 weeks to determine tolerability in the Tolerability Assessment Phase (A) prior to receiving treatment with aripiprazole IM Depot. In the Open-label Aripiprazole IM Depot Phase (B), participants received aripiprazole intramuscular (IM) Depot 400 mg injection (dosage could be adjusted to 300 mg at the investigator's discretion) monthly in the clinic for a total of 6 injections + concomitant oral aripiprazole 10-15 mg/day for the first 14 days. Participants at the investigator's discretion were eligible to continue to receive aripiprazole IM depot (400 or 300 mg) injection monthly in the Open-label Aripiprazole IM Depot Extension phase (C). Oral aripiprazole was available as rescue medication if necessary.
Period: Oral Aripirazole (Phase A)
Arm/Group | Oral Aripiprazole Tablets and Aripiprazole IM Depot Injection
Started | 19
Completed | 8
Not Completed | 11
Not completed — Sponsor discontinued study | 11
Period: Aripiprazole IM Depot Treatment Phase(B)
Arm/Group | Oral Aripiprazole Tablets and Aripiprazole IM Depot Injection
Started | 19 (Includes 8 patients from Phase A + 11 patients who entered directly into Phase B.)
Completed | 3
Not Completed | 16
Not completed — Adverse Event | 1
Not completed — Sponsor discontinued study | 13
Not completed — Subject was withdrawn by investigator | 1
Not completed — Subject withdrew consent | 1
Period: Aripiprazole IM Depot Extension Phase(C)
Arm/Group | Oral Aripiprazole Tablets and Aripiprazole IM Depot Injection
Started | 3
Completed | 0
Not Completed | 3
Not completed — Sponsor discontinued study | 3

BASELINE CHARACTERISTICS:
Population: Baseline measures are based on all enrolled participants.
Groups:
- All Participants: Patients who had no history of tolerability to oral aripiprazole received 10-15 mg/day (up to 30 mg/day) oral aripiprazole for 1 to 4 weeks to determine tolerability in the Tolerability Assessment Phase (A) prior to receiving treatment with aripiprazole IM Depot. In the Open-label Aripiprazole IM Depot Phase (B), participants received aripiprazole intramuscular (IM) Depot 400 mg injection (dosage could be adjusted to 300 mg at the investigator's discretion) monthly in the clinic for a total of 6 injections + concomitant oral aripiprazole 10-15 mg/day for the first 14 days. Participants at the investigator's discretion were eligible to continue to receive aripiprazole IM depot (400 or 300 mg) injection monthly in the Open-label Aripiprazole IM Depot Extension phase (C). Oral aripiprazole was available as rescue medication if necessary.
Arm/Group | All Participants
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.9 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 20

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Inpatient Psychiatric Hospitalization Rates
Description: The comparison of inpatient psychiatric hospitalization rates (proportion of patients with ≥1 inpatient psychiatric hospitalizations) between the retrospective period Months 4-6 (Weeks-12 to -24) while on oral standard of care antipsychotic treatment and the prospective period Phase B Months 4-6 (Weeks 12 to 24) after the switch to aripiprazole IM depot.
Time Frame: Retrospective period Months 4-6; Prospective period Months 4-6
Population: Due to the low number of enrolled patient and the sponsor's early termination of the study, the primary efficacy endpoint was not evaluated.
Groups:
- Aripiprazole IM Depot Injection: Patients who had no history of tolerability to oral aripiprazole received 10-15 mg/day (up to 30 mg/day) oral aripiprazole for 1 to 4 weeks to determine tolerability in the Tolerability Assessment Phase (A) prior to receiving treatment with aripiprazole IM Depot. In the Open-label Aripiprazole IM Depot Phase (B), participants received aripiprazole intramuscular (IM) Depot 400 mg injection (dosage could be adjusted to 300 mg at the investigator's discretion) monthly in the clinic for a total of 6 injections + concomitant oral aripiprazole 10-15 mg/day for the first 14 days. Oral aripiprazole was available as rescue medication if necessary.
- Standard of Care: Patients who received oral antipsychotic treatment as standard of care in clinical practice.
Arm/Group | Aripiprazole IM Depot Injection | Standard of Care
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change From Baseline in the Positive and Negative Syndrome Scale (PANSS) Total Score
Description: The PANSS consisted of 3 subscales with a total of 30 symptom constructs each rated on a 7-point scale where 1=absence of symptoms to 7=extremely severe symptoms. The Positive Subscale consisted of 7 positive symptom constructs with a possible subscale score of 7 to 49, the Negative Subscale consisted of 7 negative symptom constructs with a possible subscale score of 7 to 49 and the General Psychopathology Subscale consisted of 16 symptom constructs for a possible subscale score of 16 to 112. The PANSS Total Score ranged from 30 (best) to 210 (worst; indicating more severe symptoms). A Negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 24
Population: Due to the low number of enrolled patients and the sponsor's early termination of the study, this endpoint was not evaluated.
Groups:
- Aripiprazole IM Depot Injection: Patients who had no history of tolerability to oral aripiprazole received 10-15 mg/day (up to 30 mg/day) oral aripiprazole for 1 to 4 weeks to determine tolerability in the Tolerability Assessment Phase (A prior to receiving treatment with aripiprazole IM Depot. In the Open-label Aripiprazole IM Depot Phase (B), participants received aripiprazole intramuscular (IM) Depot 400 mg injection (dosage could be adjusted to 300 mg at the investigator's discretion) monthly in the clinic for a total of 6 injections + concomitant oral aripiprazole 10-15 mg/day for the first 14 days. Oral aripiprazole was available as rescue medication if necessary.
Arm/Group | Aripiprazole IM Depot Injection
Number analyzed (Participants) | 0

3. Secondary Outcome: Change From Baseline in PANSS Positive and Negative Subscale Scores
Description: The PANSS Positive Subscale consisted of 7 symptom constructs rated on a 7-point scale where 1=absence of symptoms to 7=extremely severe symptoms. The total score on the Positive Subscale ranged from 7 to 49 with a higher score indicating more severe symptoms. The PANSS Negative Subscale consisted of 7 symptom constructs rated on a 7-point scale where 1=absence of symptoms to 7=extremely severe symptoms. The total score on the Negative Subscale ranged from 7 to 49 with a higher score indicating more severe symptoms. A Negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Arm/Group | Aripiprazole IM Depot Injection
Number analyzed (Participants) | 0

4. Secondary Outcome: Clinical Global Impression of Severity (CGI-S) Score
Description: The severity of illness for each participant was rated using the CGI-S scale. The investigator answered the following question: "Considering your total clinical experience with this particular population, how mentally ill is the patient at this time?" using an 8-point scale where 0=not assessed to 7=among the most extremely ill patients.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Arm/Group | Aripiprazole IM Depot Injection
Number analyzed (Participants) | 0

5. Secondary Outcome: Clinical Global Impression of Improvement (CGI-I) Score
Description: The participant's overall improvement was rated for each participant using the CGI-I scale. The investigator rated the participant's total improvement by answering the following question: "Compared to his/her condition at baseline (prior to randomization), how much has the patient changed?" using an 8-point scale where 0=not assessed, 1=very much improved to 7=very much worse. Lower scores indicated improvement.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Arm/Group | Aripiprazole IM Depot Injection
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Groups:
- Oral Aripiprazole (Phase A): Patients who had no history of tolerability to oral aripiprazole received 10-15 mg/day (up to 30 mg/day) oral aripiprazole for 1 to 4 weeks to determine tolerability in the Tolerability Assessment Phase (A) prior to receiving treatment with aripiprazole IM Depot.
- Aripiprazole IM Depot (Phase B): In the Open-label Aripiprazole IM Depot Phase (B), participants received aripiprazole intramuscular (IM) Depot 400 mg injection (dosage could be adjusted to 300 mg at the investigator's discretion) monthly in the clinic for a total of 6 injections + concomitant oral aripiprazole 10-15 mg/day for the first 14 days. Oral aripiprazole was available as rescue medication if necessary.
- Aripiprazole IM Depot (Phase C): Participants at the investigator's discretion were eligible to continue to receive aripiprazole IM depot (400 or 300 mg) injection monthly in the Open-label Aripiprazole IM Depot Extension phase (C). Oral aripiprazole was available as rescue medication if necessary.
Arm/Group | Oral Aripiprazole (Phase A) | Aripiprazole IM Depot (Phase B) | Aripiprazole IM Depot (Phase C)
Serious Adverse Events (participants affected / at risk) | 0/19 | 1/19 | 0/3
Other Adverse Events (participants affected / at risk) | 4/19 | 10/19 | 1/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oral Aripiprazole (Phase A) (N=19) | Aripiprazole IM Depot (Phase B) (N=19) | Aripiprazole IM Depot (Phase C) (N=3)
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1 | 0
Schizophrenia (Psychiatric disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Oral Aripiprazole (Phase A) (N=19) | Aripiprazole IM Depot (Phase B) (N=19) | Aripiprazole IM Depot (Phase C) (N=3)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 3 | 3 | 0
Fatigue (General disorders) | 1 | 2 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0
Irritability (General disorders) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0
Blood glucose increased (Investigations) | 0 | 1 | 0
Blood triglycerides increased (Investigations) | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Somnolence (Nervous system disorders) | 1 | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No